CLINICAL TRIAL: NCT05624619
Title: The Diagnostic and Prognostic Value of Speckle Tracking Imaging in Septic Cardiomyopathy: a Prospective Cohort Study
Brief Title: The Diagnostic and Prognostic Value of Speckle Tracking Imaging in Septic Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: STI-01
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Sepsis; Cardiomyopathies; Echocardiography
MeSH Terms: conditions — Sepsis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to explore if STI technology, especially TMAD, plays an important role in evaluating left ventricular longitudinal systolic function and discriminating SICM in patients with sepsis. The investigators also intend to prove that TMAD may have predictive value in patients with sepsis, which is worthy of in-depth study to find strong evidence-based medical evidence for subsequent clinical practical applications.

DETAILED DESCRIPTION:
In order to explore if STI technology, especially TMAD, plays an important role in evaluating left ventricular longitudinal systolic function and discriminating SICM in patients with sepsis, the investigators intend to explore that TMAD may have predictive value in patients with sepsis, which is worthy of in-depth study to find strong evidence-based medical evidence for subsequent clinical practical applications.

ELIGIBILITY:
Inclusion Criteria:

* patients who are diagnosed as sepsis according to sepsis 3.0 criteria

Exclusion Criteria:

* patients with history of organic heart disease;
* patients with history of heart failure
* holder of cardiac implanted device;
* patients with history of atrial fibrillation;
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who are diagnosed as sepsis according to sepsis 3.0 criteria, excluding those with history of organic heart disease, heart failure, atrial fibrillation or holder of cardiac implanted device
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-18 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  28-day mortality of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Jieqiong Song, Principal Investigator — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China